CLINICAL TRIAL: NCT01159366
Title: Substudy of the Leipzig Immediate Versus Early and Late Percutaneous Coronary Intervention Trial in NSTEMI - LIPSIA-NSTEMI TRIAL
Brief Title: Incidence of Occluded Culprit Arteries and Impact of Coronary Collaterals on Outcome in Patients With NSTEMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Holger Thiele, MD, PhD, University of Leipzig
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCT00402675
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2010-07-12 (Estimated); Status verified 2010-07

CONDITIONS: NSTEMI
Keywords: myocardial infarction; coronary occlusion; myocardial revascularization; collaterals; prognosis
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; Myocardial Infarction; Coronary Occlusion | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- occluded culprit artery (Active Comparator): An occluded lesion was defined as a lesion with 100% stenosis or TIMI-flow grade 0 or 1.
  Interventions: Procedure: percutaneous coronary intervention
- non-occluded culprit artery (Active Comparator): A non-occluded lesion was defined as a lesion without 100% stenosis or TIMI-flow grade 0 or 1.
  Interventions: Procedure: percutaneous coronary intervention

INTERVENTIONS:
Procedure: percutaneous coronary intervention — early timing
  Other Names: early invasive treatment strategy in NSTEMI

SUMMARY:
It is assumed that patients with non-ST-elevation myocardial infarctions (NSTEMI) showing an infero- or posterolateral occluded culprit artery (OCA) during diagnostic angiography frequently elude standard 12-lead electrocardiogram diagnosis. In addition, coronary collaterals may have beneficial effects in patients with OCA.

DETAILED DESCRIPTION:
We examined consecutive NSTEMI patients within 48 h of symptom onset. All patients underwent early invasive angiography plus optimal medical therapy. We compared baseline characteristics, procedural findings including analysis of TIMI-flow and collaterals using the Rentrop-classification, 30-day and 6-months major adverse cardiovascular events (MACE) in patients with and without totally OCA.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 90 years,
* onset of angina pectoris at rest <24 h or crescendo angina in recent weeks with symptoms under minimal exertion or at rest lasting <24 h,
* elevated troponin T ≥0.03 µg/L and
* written informed consent.

Exclusion Criteria:

* persistent angina,
* ST-segment elevation myocardial infarction (STEMI),
* hemodynamic instability including cardiogenic shock,
* oral anticoagulation therapy,
* contraindications for glycoprotein IIb/IIIa inhibitors,
* other disease with life expectancy <6 months,
* known coagulopathy,
* pregnancy,
* other suspected causes of troponin elevation as myocarditis, secondary to hypertensive crisis, or after cardiac decompensation,
* no ability to consent, and
* participation in another study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2006-07; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
MACE | 6 months
  composite of death, reinfarction and readmission for unstable angina within 6 months after inclusion

SECONDARY OUTCOMES:
CK and CK-MB | 48 hours
  Venous blood samples were taken at admission (baseline), and every 6 h subsequently for a period of 48 h.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Schuler, MD, PhD, Study Chair — University of Leipzig
Locations (1):
- University of Leipzig, Leipzig, Germany